CLINICAL TRIAL: NCT00698555
Title: Study Comparing the Immunogenicity and Reactogenicity of Different Formulations of GSK Bio's HBV-MPL Vaccine Injected as a 0, 6 Months Schedule With That of Engerix™-B Injected as a 0, 1, 6 Months Schedule in Healthy Adults Aged 18-40 Years
Brief Title: Comparing Immunogenicity and Safety of Different Formulations of HBV-MPL Vaccine With Engerix™-B in Adults Aged 18-40 y
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/025
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBV-MPL; Recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

ARMS (6):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group B (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group C (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group D (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group E (Experimental)
  Interventions: Biological: HBV-MPL vaccine
- Group F (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine — 5 different formulations, 2-dose intramuscular injection
  Arms: Group A; Group B; Group C; Group D; Group E
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group F

SUMMARY:
This study will evaluate the immunogenicity and safety of different formulations of the candidate HBV-MPL vaccine administered according to a 2-dose schedule and compare it to that of Engerix™-B administered according to a 3-dose schedule in order to determine the optimal dose of each component of the candidate HBV-MPL vaccine when administered at 0 and 6 months

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 40 years old.
* Good physical condition as established by clinical examination and history taking at the time of entry.
* Female participants who are at risk to become pregnant will be on a contraceptive programme if necessary during the study period.
* Written informed consent obtained from the subjects

Exclusion Criteria:

* Positive titres at screening for anti-hepatitis antibodies.
* Elevated serum liver enzymes
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Any chronic drug treatment, including any treatment with immunosuppressive drugs, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous participation in any other clinical trial.
* Previous vaccination with a hepatitis B vaccine.
* Previous vaccination with an MPL containing vaccine.
* Administration of immunoglobulins in the past 6 months and during the whole study period
* Vaccination one month before and one month after each dose of the study vaccine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 1997-03; Primary Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | Month 7

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | Month 1, 2, 6 and 12
Cell mediated immunity | Month 1, 2, 6, 7 and 12
Occurrence and intensity and relationship to vaccination of solicited local and general symptoms | 4-day follow-up after vaccination
Occurrence and intensity and relationship to vaccination of unsolicited symptoms | 31-day follow-up after vaccination
Incidence of SAE | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Ghent, Belgium